CLINICAL TRIAL: NCT06369324
Title: Efficacy of Pain Neuroscience Education and Physiotherapy in Patients Diagnosed with Spondyloarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carlos Fernández-Morales, Clinical Professor, Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-04

CONDITIONS: Spondyloarthropathies; Ankylosing Spondylitis
MeSH Terms: conditions — Spondylarthropathies; Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Participants in the control group will not receive any intervention and will continue with their normal combat and flight exercise activities. They will be asked not to take medication or seek alternative treatments.
- Intervention group (Experimental): Participants in the intervention group will follow a programme of education in pain neuroscience, supervised therapeutic exercise, and an intervention based on manual therapy combined with electrical stimulation called electro-massage.
  Interventions: Other: Pain education; Other: Exercise supervised by external focus; Other: Therapy by means of electrical stimulation (electro-massage)

INTERVENTIONS:
Other: Pain education — It consisted of holding information sessions on each of the days that the subjects were scheduled for treatment. These sessions will be supported by supplementary material in the form of brochures, posters and videos which briefly explain interesting knowledge about spondyloarthropathies.
  Arms: Intervention group
Other: Exercise supervised by external focus — This therapeutic exercise involves proprioceptive training with external feedback to enhance exercise execution and promote optimal postural control, particularly for individuals with back pain. The method, based on research by Abdollahipour et al. and Chiviacowsky et al., focuses on automatic control, reducing the cognitive load during exercises and improving movement retention. The Motion Guidance Clinician Kit will be utilized, consisting of a panel and laser guide for precise cervical movement. Exercises progress in difficulty over 12 sessions, targeting cervical and lumbopelvic stabilization, flexion-extension, rotations, and lateral flexions. Sessions start with seated exercises and progress to standing, with increasing distance between laser targets to expand cervical range of motion. Thoracic and lumbar exercises involve 10 repetitions each. The entire program lasts around 20 minutes and follows Tidier recommendations for intervention.
  Arms: Intervention group
Other: Therapy by means of electrical stimulation (electro-massage) — This technique combines manual therapy (massage) with interferential current. Following a supervised therapeutic exercise program, this intervention targets the spine for 15 minutes. Using a Sonopuls 692® device, a bipolar current mode with specific frequencies is applied. The physiotherapist moistens sponges with warm water and administers the current through them while performing manual soft tissue therapy on the neck, shoulders, scapulae, thoracic, lumbar, and sacral areas. The intensity is adjusted to provide a strong but comfortable tingling sensation, without muscle twitching. The therapy sequence includes superficial stroking, deep gliding movements, trapezius kneading, muscle stretching, and deep rubbing on the thoracic and lumbar areas. The electro-massage protocol lasts 14 minutes.
  Arms: Intervention group

SUMMARY:
Spondyloarthritis, notably ankylosing spondylitis (AS), represents a chronic rheumatic condition typified by persistent back pain and stiffness. It constitutes a substantial portion of diagnoses within rheumatology units and exhibits a higher prevalence among males. Diagnosis relies upon comprehensive clinical evaluation, including patient history, physical examination, and adjunctive radiological assessments, with genetic predisposition, particularly the presence of the HLA-B27 antigen, playing a significant role.

Management strategies encompass a multidisciplinary approach, with physiotherapy emerging as a cornerstone therapeutic modality. Various exercise interventions, particularly those supervised by trained professionals, demonstrate efficacy in improving pain, stiffness, and overall functional capacity. Furthermore, patient education plays a pivotal role in enhancing treatment adherence and optimizing outcomes by aligning patient expectations with therapeutic goals.

The evolving landscape of spondyloarthritis management underscores the necessity of further research into multimodal treatment approaches, particularly in integrating novel interventions such as electrophysical agents. By elucidating the mechanisms of action and exploring their synergistic effects, clinicians can refine treatment protocols and ultimately enhance the quality of care provided to individuals living with spondyloarthritis.

DETAILED DESCRIPTION:
Spondyloarthritis or ankylosing spondylitis (AS) is a type of chronic spondyloarthropathy. According to the Spanish Society of Rheumatology (SER), spondyloarthropathies constitute a heterogeneous family of interrelated rheumatic diseases that share clinical, pathogenic, genetic, radiological, epidemiological and therapeutic response characteristics. From an epidemiological point of view, they are increasingly frequent diseases, accounting for more than 13% of patients diagnosed in rheumatology units. Specifically, international reference studies place AD as the most frequent, with an estimated incidence of 7 new cases per 100,000 inhabitants per year. It is more frequent in men than in women (in a ratio of 3:1) and the age range is between 20 and 30 years. In Extremadura the incidence is no less. According to the National Institute of Statistics (INE), there are currently 24 cases per 1000 people diagnosed with rheumatoid arthritis or AD, and 55 cases per 1000 people diagnosed with arthritis.

In terms of clinical manifestations, early symptoms include back pain and stiffness. Over time, AS can fuse vertebrae and limit movement, causing severe and constant pain. Diagnosis and follow-up of the disease is based on clinical history and physical examination. Radiological tests may also be used to complement the diagnosis. Over the years, the concept of spondyloarthropathy has evolved, and is now defined as a combination of axial spondyloarthritis (SpA), psoriatic arthritis (PsA) and inflammatory bowel disease (IBD).

With regard to the criteria according to the Assessment of Spondyloarthritis International Society (ASAS) and the latest update of the Clinical Practice Guideline for the treatment of SpA and psoriatic arthritis, within SpA the investigators find AD as the most representative pathology of this group, being the one the investigators will focus on in this research project.

The diagnosis of axial SpA requires: a) imaging evidence confirming sacroiliitis and b) at least one sign of SpA or HLA-B27 marker and two of the signs determined according to ASAS (inflammatory low back pain, arthritis, enthesitis, uveitis, dactylitis, psoriasis, Crohn's disease, good response to NSAIDs, family history of SpA, presence of HLA-B27 antigen or presence of increased C-reactive protein). In this regard, in addition to imaging and laboratory tests, the International Society for the Evaluation of SpA classification considers common clinical features as the main diagnostic axis.

Based on the latest SER review, the mechanism by which the disease occurs is still not entirely clear, although there is a genetic predisposition. Among the factors involved, the most important is the presence of the positive HLA-B27 antigen, which is present in the vast majority of patients with AD and less frequently in the rest of the diseases of the SpA group. Taking into account that only 10% of HLA-B27 antigen carriers will present with the disease, it is essential to present clinical signs to support the diagnosis.

According to the best available scientific evidence, physiotherapy is the main effective rehabilitation treatment measure for patients with SpA, and specifically for the most widespread form of the disease such as AD.

Several rehabilitation modalities exist, although, to date, there is limited consensus on a sequenced and standardised protocol. The review analysed 28 studies in which at least one intervention group received physiotherapy treatment. A total of 1926 subjects with AS were analysed, with pain, stiffness, mobility (spine and chest wall) and physical function (disease activity, ABVD and global function) being the main variables studied.

The results reported that doing physiotherapy through therapeutic exercise performed by physiotherapists is better than doing nothing. Within the exercise modalities, supervised exercise by external control or focus is showing better results in regulating pain modulatory mechanisms, also improving pain intensity, range of motion and perceived disability in subjects with spinal pathology.

On the other hand, electrophysical agents have also been routinely applied in subjects with spinal pathology, as they are inexpensive procedures with no reported adverse effects and can be easily accessible to the general population. Among these, transcutaneous electrical stimulation procedures with TENS-type currents stand out. This modality is applied via adhesive electrodes placed on the skin or on the affected nerve in question, as well as those that use medium-frequency interferential currents, showing clinical efficacy in reducing perceived pain. However, there are limited studies that apply these interventions in subjects diagnosed with AD, and as far as the authors of this project are aware, there are no clinical trials that analyse the effects of combining both interventions in a multimodal programme.

On the other hand, there are studies that demonstrate the importance of satisfaction as an influential factor in both the clinical benefits and the quality of the health care provided. If the investigators focus exclusively on the field of physiotherapy, similar benefits have been reported between those who receive an educational briefing and those who receive a standardised physiotherapy treatment without adequate information. Accurate information about the disease in question and about the stages of treatment will therefore ensure that the user's expectations are in line with reality, favouring overall satisfaction and adherence to treatment.

In this context, there has been a growing interest in analysing multimodal physiotherapy programmes in the approach to chronic musculoskeletal pathology.

ELIGIBILITY:
Inclusion Criteria:

* Adults (men and women) over 18-65 years of age.
* Diagnosed with ankylosing spondylitis by a rheumatologist.

Exclusion Criteria:

* Sample subjects with spinal surgery in the last 12 months were excluded.
* Subjects with mild/moderate cognitive impairment (score ≥24 in the Spanish validated version for general older adults of the Mini-Mental State Examination) (Lobo A, Saz P, Marcos G et al. Revalidation and standardisation .
* Finally, those with pharmacological treatment that could generate vestibular or balance disturbances at the time of assessment and treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4 weeks.
  Numeric Pain Rating Scale (NPRS) is a 11-point numeric rating scale, where 0 denotes "no pain" and 10 denotes "the maximum bearable pain". The minimum clinically important difference (MCID) for this tool has been established at 1.5 points and the minimum detectable change (MDC) at 2.6 points, in individuals with neck pain. The NPRS is a valid scale with moderate test-retest reliability in this population (Intraclass Coefficient Correlation (ICC): 0.76, 95% CI 0.58 to 0.93).
Cervical and Lumbar Joint Position Sense Error | 4 weeks.
  This test consists of a visual measurement of the error when moving the head to the initial neutral position after active cervical rotation, or when performing lumbar flexion or extension and returning to a neutral position.
Cervical Range of Motion (CRoM) | 4 weeks.
  For the evaluation of CROM, a conventional EnrafNonius® two-branch goniometer was used. Subjects were placed in a seated position on a stool, with a neutral neck and head position. The range of active cervical mobility presented by the patients was measured in reference to the three planes of the space. In the sagittal plane, the degrees of mobility to flexion and extension were measured, in the frontal plane the right and left inclinations, and in the transverse plane both rotations.
Pressure Pain Threshold (PPT) | 4 weeks.
  A mechanical pressure Fisher algometer (Force Dial model FDK 40) with a 1 cm² area contact head was used to measure the pressure pain threshold. The reliability of pressure algometry has been found to be high [intraclass correlation coefficient = 0.91 (95% confidence interval, 0.82-0.97)]. With the participant in supine, the pressure pain threshold of the the myofascial trigger point nº2 of the upper trapezius muscle according to Travell and Simons and the central trigger point of the sternocleidomastoid muscle was bilaterally evaluated. Also, in sitting position the pressure pain threshold of the myofascial trigger point of the scapula elevator muscle was bilaterally evaluated. The minimal clinically important difference (MCDI) is 1.2 Kg/cm2.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 4 weeks.
  Is a questionnaire used to assess disease activity and severity in individuals with ankylosing spondylitis, focusing on symptoms such as pain, stiffness, and fatigue. The minimum score is 0 and the maximum score is 60. Higher scores indicate a worse outcome.
Bath Ankylosing Spondylitis Motility Index (BASMI) | 4 weeks.
  The Bath Ankylosing Spondylitis Motility Index (BASMI) explores the mobility of the spine and hips and includes the Schober test to indicate the degree of mobility of the lumbar tract. The minimum score is 0 and the maximum score is 10. Higher scores indicate a worse outcome.
Bath Ankylosing Spondylitis Functional Index (BASFI). | 4 weeks.
  The Bath Ankylosing Spondylitis Functional Index (BASFI) is a questionnaire used to evaluate the functional ability and physical functioning of individuals with ankylosing spondylitis. It assesses aspects such as activities of daily living, mobility, and overall function, providing a measure of disease impact on a person's life. The minimum score is 0 and the maximum score is 100. Higher scores indicate a worse outcome.
Kinesophobia | 4 weeks.
  The Spanish version of the TSK-11 was used to measure fear of movement. Higher scores indicate greater fear-avoidance behaviors. The TSK-11 has demonstrated acceptable internal consistency and validity.
Catastrophizing Pain | 4 weeks.
  The Pain Catastrophizing Scale (PCS) is a self-administered scale of 13 items and one of the most used to assess catastrophism of pain. The subjects take their past painful experiences as a reference and indicate the degree to which they experienced each of the 13 thoughts or feelings on a 5-point Líkert scale ranging from 0 (never) to 4 (always). The theoretical range of the instrument is between 13 and 62, indicating low scores, little catastrophism, and high values, high catastrophism.
Fear-Avoidance Beliefs Questionnaire (FABQ) | 4 weeks.
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a self-report measure designed to assess beliefs and attitudes related to fear of movement and avoidance behavior in individuals with musculoskeletal pain, particularly low back pain. It evaluates the extent to which individuals perceive physical activity as harmful and the degree to which they avoid certain activities due to fear of exacerbating their pain. The minimum score is 0 and the maximum score is 96. Higher scores indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo-Antúnez, Ph.D, Study Director — University of Extremadura
Locations (1):
- Faculty of Medicine and Health Sciences, Badajoz, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albornoz-Cabello M, Barrios-Quinta CJ, Espejo-Antunez L, Escobio-Prieto I, Casuso-Holgado MJ, Heredia-Rizo AM. Immediate clinical benefits of combining therapeutic exercise and interferential therapy in adults with chronic neck pain: a randomized controlled trial. Eur J Phys Rehabil Med. 2021 Oct;57(5):767-774. doi: 10.23736/S1973-9087.21.06688-0. Epub 2021 Mar 24. PMID 33759439
- [Background] Albornoz-Cabello M, Sanchez-Santos JA, Melero-Suarez R, Heredia-Rizo AM, Espejo-Antunez L. Effects of Adding Interferential Therapy Electro-Massage to Usual Care after Surgery in Subacromial Pain Syndrome: A Randomized Clinical Trial. J Clin Med. 2019 Feb 2;8(2):175. doi: 10.3390/jcm8020175. PMID 30717426
- [Background] Dougados M, van der Linden S, Juhlin R, Huitfeldt B, Amor B, Calin A, Cats A, Dijkmans B, Olivieri I, Pasero G, et al. The European Spondylarthropathy Study Group preliminary criteria for the classification of spondylarthropathy. Arthritis Rheum. 1991 Oct;34(10):1218-27. doi: 10.1002/art.1780341003. PMID 1930310
- [Background] Frost H, Lamb SE, Doll HA, Carver PT, Stewart-Brown S. Randomised controlled trial of physiotherapy compared with advice for low back pain. BMJ. 2004 Sep 25;329(7468):708. doi: 10.1136/bmj.38216.868808.7C. Epub 2004 Sep 17. PMID 15377573
- [Background] Lara-Palomo IC, Aguilar-Ferrandiz ME, Mataran-Penarrocha GA, Saavedra-Hernandez M, Granero-Molina J, Fernandez-Sola C, Castro-Sanchez AM. Short-term effects of interferential current electro-massage in adults with chronic non-specific low back pain: a randomized controlled trial. Clin Rehabil. 2013 May;27(5):439-49. doi: 10.1177/0269215512460780. Epub 2012 Oct 3. PMID 23035006
- [Background] Navarro-Compan V, Sepriano A, El-Zorkany B, van der Heijde D. Axial spondyloarthritis. Ann Rheum Dis. 2021 Dec;80(12):1511-1521. doi: 10.1136/annrheumdis-2021-221035. Epub 2021 Oct 6. PMID 34615639
- [Background] Rudwaleit M, van der Heijde D, Landewe R, Akkoc N, Brandt J, Chou CT, Dougados M, Huang F, Gu J, Kirazli Y, Van den Bosch F, Olivieri I, Roussou E, Scarpato S, Sorensen IJ, Valle-Onate R, Weber U, Wei J, Sieper J. The Assessment of SpondyloArthritis International Society classification criteria for peripheral spondyloarthritis and for spondyloarthritis in general. Ann Rheum Dis. 2011 Jan;70(1):25-31. doi: 10.1136/ard.2010.133645. Epub 2010 Nov 24. PMID 21109520
- [Background] Sharan D, Rajkumar JS. Physiotherapy for Ankylosing Spondylitis: Systematic Review and a Proposed Rehabilitation Protocol. Curr Rheumatol Rev. 2017;13(2):121-125. doi: 10.2174/1573397112666161025112750. PMID 27784233
- [Background] van der Linden S, Valkenburg HA, Cats A. Evaluation of diagnostic criteria for ankylosing spondylitis. A proposal for modification of the New York criteria. Arthritis Rheum. 1984 Apr;27(4):361-8. doi: 10.1002/art.1780270401. PMID 6231933
- [Background] Zao A, Cantista P. The role of land and aquatic exercise in ankylosing spondylitis: a systematic review. Rheumatol Int. 2017 Dec;37(12):1979-1990. doi: 10.1007/s00296-017-3829-8. Epub 2017 Oct 5. PMID 28983663